CLINICAL TRIAL: NCT05549947
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacokinetics of SHR-1819 Injection in Adults With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Study of SHR-1819 Injection in Adult Patients With Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHR-1819-201
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A：SHR-1819 (Experimental)
  Interventions: Drug: SHR1819
- Treatment group B：SHR-1819 (Experimental)
  Interventions: Drug: SHR1819
- Treatment group C：SHR-1819 (Experimental)
  Interventions: Drug: SHR1819
- Treatment group D：placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR1819 — Treatment group A：SHR-1819 injection dose 1， Treatment group B：SHR-1819 injection dose 2， Treatment group C：SHR-1819 injection dose 3，
  Arms: Treatment group A：SHR-1819; Treatment group B：SHR-1819; Treatment group C：SHR-1819
Drug: Placebo — Treatment group D：placebo
  Arms: Treatment group D：placebo

SUMMARY:
This trial was designed to evaluate the efficacy and safety of SHR-1819 injection in patients with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign informed consent forms prior to the commencement of any proceedings related to the study, are able to communicate smoothly with the investigator, understand and are willing to complete the study in strict compliance with the requirements of this clinical research protocol；
2. Age 18 to 75 years old (inclusive) at the time of signing the informed consent form, regardless of gender;
3. Have atopic dermatitis at the time of screening (according to the 2014 American College of Dermatology Guidelines) and have a course of at least 1 year before screening;
4. At the screening and baseline periods, EASI ≥ 16, IGA ≥3, BSA ≥ 10 %
5. The average daily peak pruritus (itch) numerical evaluation scale (P-NRS) score for the first 7 days of randomization ≥4 points (at least 4 days of daily peak pruritus P-NRS scores need to be collected);
6. According to the investigators, topical TCS treatment was poor or intolerant within 6 months prior to screening

Exclusion Criteria:

1. Pregnant or lactating women
2. Major surgeries are planned for the duration of the study
3. History of previous atopic corneal conjunctivitis involving the cornea
4. History of clinically significant diseases (e.g., circulatory system abnormalities, endocrine system abnormalities, neurological disorders, hematologic disorders, immune system disorders, psychiatric disorders, and metabolic instability) that the researcher believes that participation in the study poses a risk to the safety of the subject or that the disease/illness worsens during the study period will affect the effectiveness or safety analysis.
5. Subjects have had or are currently clinically significant diseases or abnormalities
6. Screening for people with a history of heavy alcohol consumption or substance abuse in the 3 months prior to screening
7. The drug has been used in the previous 6 months
8. Screening of subjects with malignancy within the first 5 years (except completely cured cervical cancer in situ and non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma)
9. Other comorbid (or co-occurring) skin disorders may be affected in the study evaluation
10. Any cause that the researchers believe would prevent the participants from participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
At 16 weeks, the proportion of subjects who achieved eczema area and severity index (EASI) -75 (EASI score decreased ≥75% from baseline) | up to 16 weeks
  EASI sore use EASI scale

SECONDARY OUTCOMES:
At week 16, the proportion of participants with an overall investigator assessment (IGA) score of 0 or 1 (0-4 scale) and a decrease of ≥2 points from baseline | up to 16 weeks]
  The overall degree of improvement was assessed using the IGA scale
At week 16, the proportion of subjects whose IGA score decreased from baseline by ≥2 points; | up to 16 weeks
  The overall degree of improvement was assessed using the IGA scale
At week 16, the proportion of subjects who achieved EASI-90 (EASI score ≥90% lower than baseline); | up to 16 weeks
  The extent of area is assessed using the EASI scale
At week 16, the percentage of subjects who achieved EASI-50 (EASI score ≥50% lower than baseline); | up to 16 weeks
  The extent of area is assessed using the EASI scale
At week 16, the weekly average of the daily peak itching (itch) digital evaluation scale (P-NRS) decreased from baseline by ≥4 points | up to 16 weeks
  The extent of pruritus is assessed using the P-NRS scale
At week 16, EASI is the percentage change from baseline and change; | up to 16 weeks
  The extent of area is assessed using the EASI scale
At week 16, the atopic dermatitis score (SCORAD) was the percentage change from baseline and change | up to 16 weeks
  The extent of lesions and pruritus is assessed using the SCORAD scale
At week 16, atopic dermatitis affects the body surface area (BSA) as a percentage of the baseline change and change | up to 16 weeks
  The BSA scale was used to assess improvement in lesion area
At week 16, the Dermatological Quality of Life Scale (DLQI) score was a percentage change from baseline and change. | up to 16 weeks
  The quality of Life is assessed using the DLQI scale
The incidence of adverse events ranged from the first dose to 24 weeks | From the beginning of administration to the 24th week
  Assess the post-medication safety of subjects from the first dose to the time they exit the group
The concentration of SHR-1819 in serum :Cmax | From the beginning of administration to the 24th week
  The concentration of SHR-1819 in plasma will be determined
The time of metabolism of the drug in the serum | From the beginning of administration to the 24th week
  The concentration of SHR-1819 in plasma will be determined
The concentration of SHR-1819 in serum :AUC | From the beginning of administration to the 24th week
  The concentration of SHR-1819 in plasma will be determined
Changes in the level of TARC in the serum | From the beginning of administration to the 24th week
  Changes in the level of biomarkers in serum
Changes in the level of CCL17 in the serum | From the beginning of administration to the 24th week
  Changes in the level of biomarkers in serum
Changes in the level of IgE in the serum | From the beginning of administration to the 24th week
  Changes in the level of biomarkers in serum
Immunogenic endpoint: evaluate the incidence and timing of ADA positivity for SHR-1819 | From the beginning of administration to the 24th week
  Changes in the level of immunogenicity in the body

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Sub-Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided